CLINICAL TRIAL: NCT04819035
Title: Post Market Clinical Utility of ESId (MDW Hematology Parameter) for Early Sepsis Detection in the Emergency Department (US Hospitals) - Indiana University Hospital
Brief Title: Sepsis Post Market Clinical Utility Simple Endpoint Study - Indiana University Hospital
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C54020
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Sepsis; Adult Disease; Severe Sepsis; Emergency Department
MeSH Terms: conditions — Sepsis; Disease; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CBC-Diff Monocyte Volume Width Distribution: Monocyte Volume Width Distribution (MDW) is part of the CBC with Differential
  Interventions: Diagnostic Test: CBC-DIFF Monocyte Volume Width Distribution (MDW)

INTERVENTIONS:
Diagnostic Test: CBC-DIFF Monocyte Volume Width Distribution (MDW) — MDW measurement will be used to detect sepsis. Results will not be used to manage patients.

SUMMARY:
The purpose of this study is to demonstrate that addition of the Monocyte Width Distribution (MDW) parameter to current standard of care improves a clinician's ability to recognize sepsis in the Emergency Department, resulting in earlier decision to administer antibiotics from time of ED presentation for sepsis patients (simulated primary endpoint), with concomitant reductions in length of stay and in-hospital mortality for those patients (secondary endpoints).

DETAILED DESCRIPTION:
The objective of this study is to develop a method for identifying sepsis patients from electronic health records (EHR) based on Sepsis-2 criteria. Sepsis patients will be identified using a Sepsis Definition which includes meeting SIRS score of ≥2 within 12 hours of ED presentation and any microbial testing ordered within 24 hours of ED presentation. The patient will be enrolled if it meets the Sepsis Definition and additional EMR data elements will be extracted to complete case report form. Furthermore, objectives include to confirm the clinical validity and performance of MDW in a control population of sepsis patients where MDW is measured but not reported to physicians. This study is an observational study which will simulate the decision impact of MDW on sepsis identification and patient management

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 to 89 years)
* All race and ethnicities
* Presenting to the emergency department with suspicion of infection
* Whose assessment includes a CBC with differential
* Meets EMR Sepsis Definition

Exclusion Criteria:

* Pregnancy
* Prisoners
* Transfers from other ED
* Previously enrolled

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to the ED where a CBC-Diff has been ordered by standard of care
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Potential reduction of Time to Antibiotics Ordered and Administered | Within 12 hours from presentation to the emergency department
  Monocyte Distribution Width's [MDW] ability to reduce time to first antibiotics ordered by physician (decision to treat) and first antibiotics administered via a simulation

SECONDARY OUTCOMES:
Performance | Within 12 hours from presentation to the emergency department
  Monocyte Distribution Width's [MDW] ability to identify Sepsis vs Non-Sepsis when using a Sepsis electronic medical record definition using AUC (Area Under The Curve) ROC (Receiver Operating Characteristics) curve.

OTHER OUTCOMES:
Health & Economic Benefits for Hospital Stay - Simulated | Within 12 hours from presentation to the emergency department
  Monocyte Distribution Width's [MDW] ability to reduce length of hospital stay by earlier detection of sepsis by using AUC (Area Under The Curve) ROC (Receiver Operating Characteristics) curve.
Health & Economic Benefits for Intensive Care Unit Stay - Simulated | Within 12 hours from presentation to the emergency department
  Monocyte Distribution Width's [MDW] ability to reduce length of intensive care unit stay by earlier detection of sepsis by using AUC (Area Under The Curve) ROC (Receiver Operating Characteristics) curve.
Health & Economic Benefits for Mortality - Simulated | Within 12 hours from presentation to the emergency department
  Monocyte Distribution Width's [MDW] ability to reduce in-house mortality by earlier detection of sepsis by using AUC (Area Under The Curve) ROC (Receiver Operating Characteristics) curve.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Czader, MD, Principal Investigator — Indiana University Health
Locations (1):
- Indiana University Methodist Hospital, Indianapolis, Indiana, United States